CLINICAL TRIAL: NCT07225465
Title: The Evaluation of Two Response Thresholds to Continuous Ketone Monitoring Information Minimising Ketosis in People With Type 1 Diabetes Treated With Dapagliflozin
Brief Title: Evaluating Safe Ketone Thresholds To Minimise Ketosis in People With Type 1 Diabetes Using Dapagliflozin
Acronym: KETO-TRACK
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: Baker Heart and Diabetes Institute (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Melbourne (Other); Melbourne Health (Other); Austin Health (Other Government)
Responsible Party: Principal Investigator, David O'Neal, Coordinating Principal Investigator, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 235/25; 1U01DK143330-01 (NIH)
Record Dates: First submitted 2025-11-02; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Ketosis; Dapagliflozin; Type 1 Diabetes; Dual Glucose and Ketone Monitor; SGLT2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Ketosis | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual glucose and ketone (DGK) sensor threshold 1.0mmol/L (Active Comparator): The DGK will be set with threshold alarms activated at 1.0mmol/L for participant response to ketosis
  Interventions: Drug: FORXIGA
- Dual glucose and ketone (DGK) sensor threshold 1.5mmol/L (Active Comparator): The DGK will be set with threshold alarms activated at 1.5mmol/L for participant response to ketosis
  Interventions: Drug: FORXIGA

INTERVENTIONS:
Drug: FORXIGA — All participants will take FORXIGA (Dapagliflozin) orally at a dose of 10mg/day for 12 weeks

SUMMARY:
Sodium glucose cotransporter 2 (SGLT2) inhibitors are a type of medicine that help the kidneys get rid of extra sugar in the blood through urine. In people with type 2 diabetes (T2D), these medications help lower blood sugar levels, help people lose weight and improve heart and kidney health.

SGLT2 inhibitors are mainly used in T2D, however some studies show they might also help people with type 1 diabetes (T1D). The same health benefits observed in people with T2D the investigators anticipate may help those with T1D. Currently, there is a safety concern that people with T1D using these medicines can raise the risk of diabetic ketoacidosis (DKA). DKA occurs when the body doesn't have enough insulin (a hormone made in the pancreas that helps your body use sugar (glucose) for energy), it starts to break down fats as a source of energy. This breakdown of fats produces ketones. Very high levels of ketones in the blood can make the blood acidic (toxic) and lead to DKA. If not treated in time, this can make the person living with T1D very ill and can be life-threatening. Because of this risk, health agencies like the FDA in the U.S., and the TGA in Australia have not approved use of SGLT2 inhibitors for people with T1D.

Still, some experts believe SGLT2 inhibitors may safely be used alongside insulin in T1D if DKA risk is carefully managed. This might be possible with early detection and treatment of rising ketone levels. One approach is using continuous ketone monitors, which track ketone levels in real time and can alert users early. People would also need proper education on what to do if ketone levels start rising.

To date, there's no official agreement on the exact ketone level that should trigger action. Some suggest action when ketone levels reach 1.0 or 1.5 mmol/L. A lower limit like 1.0 mmol/L may be safer, but it could also lead to too many alarms and extra stress, or unnecessary eating to bring ketones down.

Therefore, the aim of this study is to assess if initiating responses to elevated ketone levels at a threshold of 1.0 mmol/L, compared to a threshold of 1.5 mmol/L, will reduce the risk of DKA in people with T1D using Dapagliflozin.

The investigators will recruit 115 adults with T1D and provide Dapagliflozin (SGLT2 inhibitor) and continuous glucose and ketone monitoring (DGK) devices. Participants will be randomly assigned to two groups. Group 1 will wear a DGK with alarms set at ketone level of 1.0 mmol/L and receive education about taking action when ketone levels are ≥1.0 mmol/L. Group 2 will wear a DGK with alarms set at ketone level of 1.5 mmol/L and receive education about taking action when ketone levels are ≥1.5 mmol/L. Participants will be assessed for time spent with critically high ketone levels, incidence of DKA, glucose and person reported outcomes.

Findings from this study will provide real life data and clinical evidence to help guide safe use of SGLT2 inhibitors in people with T1D by informing protocols for monitoring and managing associated DKA risks.

DETAILED DESCRIPTION:
Sodium glucose cotransporter 2 (SGLT2) is responsible for approximately 90% of glucose re-absorption in the renal proximal tubules, so SGLT2 inhibition results in significant excretion of glucose in the urine. SGLT2 inhibition may play a key role in the prevention and management of the cardiovascular-kidney-metabolic (CKM) syndrome as this class of agent has been shown to benefit glucose levels (reducing HbA1c, and glycaemic variability without increasing severe or total hypoglycaemia), reduce heart failure, improve weight control, reduce cardiovascular mortality, and provide reno-protection in people with diabetes thereby addressing some of the fundamental issues contributing to the syndrome. While most data pertain to agents which inhibit SGLT2 in people with T2D, SGLT2 inhibition also has the potential to substantially benefit glucose control, weight management, and reduce complication development including that of the CKM syndrome in people with T1D. Dapagliflozin is a SGLT2 inhibitor. Data available in adults with T1D indicate that Dapagliflozin improves glucose control without increasing hypoglycaemia and reduces glycaemic variability. In addition, there are improvements in body weight and blood pressure. There is also substantial evidence in people with T2D that Dapagliflozin lowers mortality from cardiovascular causes and hospitalisations for heart failure. In terms of reno-protective effects, Dapagliflozin was demonstrated to slow down decline in renal function, reduce rates of renal failure and death from renal causes in T2D.These cardiorenal benefits may extend to people with T1D.

While SGLT2 inhibitors as adjunctive therapy to insulin may benefit people with T1D, in general their use has been associated with a significantly increased risk of diabetic ketoacidosis (DKA) which may occur in the absence of hyperglycaemia. DKA represents a life-threatening acute emergency of T1D, which occurs when insulin deficiency leads to lipolysis and accumulation of ketones, resulting in metabolic acidosis. It requires prompt identification and action, and delays in management are associated with an increase in mortality. For example, the pooled analysis of DEPICT-1 and DEPICT-2 participants showed that over 52 weeks of treatment, the incidence of adjudicated DKA was numerically higher with Dapagliflozin 5 mg/day or 10 mg/day than with placebo (4.0% and 3.5% vs. 1.1%). Therefore, SGLT2 inhibitors in general have failed to receive approval in the USA (FDA) and Australia (TGA) for use to control glucose levels in people with T1D due to an unacceptable increase in DKA. It is possible that SGLT2 inhibitor therapy may be viable in people with T1D if an intervention is able to shift the risk-benefit balance in favour of benefit e.g. if the risk of DKA could be recognized and addressed in a timely manner. The early recognition of impending DKA is of critical importance. However, symptoms of ketosis which include nausea, vomiting, fatigue, loss of appetite, malaise, weakness, and tachypnoea appear late and those associated with dehydration may be absent in the setting of normoglycaemia. Therefore, timely ketone measurement represents a cornerstone of management allowing therapeutic measures to be initiated.

A continuous ketone sensor (CKS) would address many of the shortcomings associated with current standard-of-care blood ketone testing using a handheld meter. Ketones can be quantified in interstitial fluid using a similar approach to that taken with widely commercially used continuous glucose monitor (CGM), using an enzymatic reaction. While feasibility of CKS devices has previously been demonstrated, the optimum thresholds for alerts, balancing the burden of alarms vs. timely intervention, have yet to be determined. Preliminary at home CKS data provided by Abbott indicate free-living people with T1D who are not using SGLTi spend <1% of the time with ketone levels >1.0mmol/L. Ketone levels in free-living with T1D using SGLT2 inhibitors remains unknown. To provide insights into appropriate ketone thresholds for alerts a literature search was undertaken in May 2024.

Studies included were published between January 2000 and April 2024 involving those aged ≥16 years of age which described capillary β-OHB levels in relation to suspected DKA and which reported sensitivity, specificity, negative predictive value, or positive predictive value. Eight of the 11 studies provided capillary β-OHB levels that excluded DKA; these ranged from 0.7 to ≥3.0 mmol/L 13-23 and the most recommended cut-off level was 1.0 mmol/L (n=3) followed by 1.5 mmol/L (n=2). The β-OHB cut-offs for the diagnosis of DKA ranged from 1.8 mmol/L to 3.5 mmol/L, with 3.0 mmol/L being most proposed by five of the studies. The investigators therefore concluded that capillary β-OHB cut off values of <1.0 mmol/L and <1.5 mmol/L exclude DKA. The investigators also conclude that a capillary β-OHB level ≥3.0 mmol/L exhibited high sensitivity and specificity in detecting DKA with levels between 1.5 mmol/L and 3.0 mmol/L representing a transition range with increasing risk.

The investigators propose that to pre-empt DKA in people with T1D using SGLTi that responses to CKS data could be initiated at levels of either 1.0mmol/L or 1.5mmol/L with alerts aligned accordingly. The lower alert may provide an additional safety margin though could come at the cost of a greater number of alarms and carbohydrates eaten that may not have necessarily been required. The investigators also suggest that there may be high DKA-risk subgroups (female sex, lower baseline body mass index (BMI), β-hydroxybutyrate levels pre-treatment, use of an insulin pump, and lower insulin requirements at baseline with dose reductions required post SGLT inhibitor commencement to avoid hypoglycaemia) who may benefit from the lower alarm thresholds facilitating earlier intervention. Finally, the risk for DKA may vary according to illness, fasting and high intensity exercise requiring alerts to be adjusted according to circumstances. However, data are required to inform protocols.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 24 and 85 years of age inclusive (66% 24Y to 65Y; and 33% >65Y to 85Y)
* Diagnosed with T1D (made on clinical criteria) for at least 1 year
* Insulin regimen either on MDI or insulin pump with at least 40% in one mode
* Minimum total daily insulin dose 0.4 Units per kg / day (can be on insulin pump or MDI);
* HbA1c <10% (86mmol/ mol)
* Minimum daily carbohydrate intake of 100g
* Willing to adhere to the study protocol
* Ability to perform high-intensity exercise (specific to the exercise sub-study)

Exclusion Criteria:

* Pregnancy or planned pregnancy
* eGFR <30ml/min/1.73m2
* History of DKA in the last 12 months
* Use of low carbohydrate diet (<100g/day)
* Diabetic gastroparesis
* Tape allergy
* Heavy alcohol use (15 standard drinks per week or binge drinking)
* Use of SGLT inhibitor in the last month
* Medications increasing the risk of DKA e.g. steroids, anorectic agents (eg phentermine, naltrexone HCl/bupropion HCl, and GLP 1 agonists).
* Major medical or psychiatric illness that in the opinion of the investigator would interfere with protocol adherence or impact participant safety.

Ages: 24 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percent time spent with interstitial ketones ≥3.0mmol/L (Main Study) | Commencement to end of study (12 weeks)
  Percent of time spent with interstitial ketone levels ≥3.0mmol/L on dual glucose / ketone monitoring device during 12-weeks of taking Dapagliflozin
Percent of time spent with interstitial ketones ≥3.0mmol/L during exercise (Exercise Study) | Weeks 4 to12
  Percent of time spent with interstitial ketones ≥3.0mmol/L on dual glucose / ketone monitoring device from start of exercise to 12 hours post-commencement of exercise

SECONDARY OUTCOMES:
Percent of time with ketone levels in different ranges | Commencement to end of study (12 weeks)
  Percent time with interstitial ketone levels of:
  1. >0.6 mmol/L
  2. >1.0 mmol/L
  3. >1.5mmol/L
Mean interstitial ketone levels | Commencement to end of study (12 weeks)
  Average if ketone levels measured by dual glucose / ketone monitor device over 12 weeks
Incidence of diabetic ketoacidosis (DKA) | Commencement to end of study (12 weeks)
  Number of DKA events
Change in HbA1c | Week 0 and Week 12 from study commencement
  Difference in HbA1c (mmol/mol) between baseline and study end
CGM metrics | Commencement to end of study (12 weeks)
  Standardised consensus CGM metrics (% times in prespecified ranges, mean glucose, and CV) over 12 weeks
Change in weight | Week 0 and Week 12 from study commencement
  Change in weight (kg) from baseline to study end
Change in BMI | Week 0 and Week 12 from study commencement
  Change in BMI (kg/m2) from baseline to study end
Change in treatment satisfaction using Diabetes Medication System Rating Questionnaire - Short form | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 20 items. Items are scored on a scale from 0 to 3-4. Higher scores mean better outcome
Change in Gold score | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 1 item. Item is scored on a scale from 1 to 7. Higher scores mean worse outcome
Change in Pittsburgh Sleep Quality Index | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 19 items. Items are scored on a scale from 0 to 3. Higher scores mean worse outcome
Change in PROMIS Fatigue - Short form | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 4 items. Items are scored on a scale from 1 to 5. Higher scores mean worse outcome
Change in EQ-5D-5L | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 6 items. Items are scored on a scale from 1 to 5. Higher scores mean worse outcome
Change in Problem Areas in Diabetes - Short form | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 5 items. Items are scored on a scale from 0 to 4. Higher scores mean worse outcome
Change in WHO-5 Well-being index | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 5 items. Items are scored on a scale from 0 to 5. Higher scores mean better outcome
Change in Hypoglycaemia Fear Survey - Short Form | Week 0 and Week 12 from study commencement
  Change in questionnaire scores from baseline to study end. Questionnaire contains 11items. Items are scored on a scale from 0 to 4. Higher scores mean worse outcome
Treatment satisfaction with ketone sensor using Study specific questions regarding treatment satisfaction | Week 12 from study commencement (study end)
  Questionnaire contains 10 items. Items are scored on a scale from 1 to 5. Higher scores mean better outcome
Ketone sensor usability with System Usability Scale | Week 12 from study commencement (study end)
  Questionnaire contains 10 items. Items are scored on a scale from 1-5. Higher scores mean better outcome
Treatment satisfaction and ketone sensor usability with User Experience Questionnaire | Week 12 from study commencement (study end)
  Change in questionnaire scores from baseline to study end. Questionnaire contains 26 items. Items are scored on a scale from 1 to 7. Higher scores mean better outcome
Lived experience of a using DGK system during Dapagliflozin treatment | Week 12 from study commencement (study end)
  Thematic analysis of interviews exploring lived experience of a using DGK system during Dapagliflozin treatment

OTHER OUTCOMES:
Percent time of sensor wear | Commencement to end of study (12 weeks)
  Percentage of time dual glucose/ketone sensor is worn during the 12 weeks of the study
Incidence of sensor- related skin infections | Commencement to end of study (12 weeks)
  Number of skin infections at site of sensor insertion
Mean duration of sensor survival before replacement | Commencement to end of study (12 weeks)
  Number of days dual glucose/ketone sensor is working for before needing replacement
Difference between blood and interstitial ketones values | Commencement to end of study (12 weeks)
  Difference between ketone readings from the dual ketone/glucose sensor (study sensor) and fingerprick blood ketone test (standard of care)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Baker Heart and Diabetes Institute, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No